CLINICAL TRIAL: NCT07027111
Title: A Phase 2, Open-label Study to Evaluate the Safety, Tolerability, and Efficacy of Intravenous NVG-2089 in Participants With Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Brief Title: Safety, Tolerability, and Efficacy of NVG-2089 in Participants With CIDP
Acronym: INVGOR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nuvig Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NVG-2089-201; 2024-515386-34-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-02; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Experienced (Experimental)
  Interventions: Drug: NVG-2089
- Treatment Naive (Experimental)
  Interventions: Drug: NVG-2089

INTERVENTIONS:
Drug: NVG-2089 — Study drug

SUMMARY:
The purpose of the study is to evaluate the safety of NVG-2089 and to evaluate how well patients respond to this investigational treatment. NVG-2089 is a new drug that is being developed for treating patients with CIDP. NVG-2089 is designed to mimic the effects of a protein called IVIg. NVG-2089 is designed to potentially help the immune system by attaching (binding) to certain receptors in the body and activating them, which helps reduce inflammation and supports how the immune system works.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years of age at the time of signing the ICF.
* Diagnosed with CIDP or Possible CIDP according to criteria of the EAN/PNS 2021 (Van den Bergh, 2021). (Diagnosis is to be confirmed by an independent adjudication committee; refer to Section 8.1.1).
* Must have an adjusted INCAT score as follows:

  1. Treatment-naïve participants: ≥2 at screening
  2. Treatment-experienced participants: 2-7 at screening Note: A score of 2 should be exclusively from leg disability component of adjusted INCAT. For participants with an adjusted INCAT score of ≥3 (and up to 7 for treatment-experienced; no upper limit for treatment-naïve) at study entry, there are no specific requirements for arm or leg scores.
* Treatment-experienced participants: Participants who were treated with IVIg/SCIg at the time of screening must have documented evidence within 24 months of screening of:

  1. Clinically meaningful deterioration on treatment interruption or dose reduction of standard of care (SOC) therapy, determined by clinical examination documented in the medical records. Clinically meaningful deterioration is defined as one of the following: ≥1-point increase in adjusted INCAT score, decrease in I-RODS total score ≥4 points, decrease in MRC Sum score ≥3, grip strength worsening of ≥8 kPa (in either hand), or an equivalent deterioration based on information from medical records and at the investigator's judgement.

     OR
  2. Improvement in CIDP symptoms with SOC therapy based on information in medical records and at the investigator's judgement. In assessing the history of response to IVIg/SCIg, the investigator should account for prior treatment (type, dose regimen, duration), pattern of response or non-response to treatment.
* a. Treatment-naïve participants: No prior treatment with IVIg and/or SCIg and/or corticosteroids and/or investigational therapies for CIDP.

OR b. Treatment-experienced participants: On stable dose of IVIg or SCIg with no disease exacerbations for 8 weeks prior to screening. Participants must be willing to discontinue IVIg or SCIg at least 3 weeks (±1 week) prior to dosing with the study drug. Participants on IVIg must be on maintenance dose of 0.4 to 1 g/kg every 2 to 6 weeks per EAN/PNS recommendation. Participants on SCIg should not exceed the dose of 0.4 g/kg per week.

Exclusion Criteria:

* Pure sensory or distal CIDP variants (EAN/PNS definition)
* History of being non-responder or loss of response to IVIg or SCIg per Investigator's determination. In assessing the history of response or loss of response to IVIg/SCIg, the investigator should account for prior treatment (type, dose regimen, duration), pattern of response or non-response to treatment. Note, participants who are on IVIg but relapsed on SCIg will be allowed to enter the study.
* Polyneuropathy of other causes, including the following: multifocal motor neuropathy; polyneuropathy associated with anti-myelin associated glycoprotein (MAG) antibodies, polyneuropathy associated with IgM monoclonal gammopathy; hereditary demyelinating neuropathy; polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin change syndromes (POEMS); lumbosacral radiculoplexus neuropathy; polyneuropathy most likely due to diabetes mellitus; polyneuropathy most likely due to systemic illnesses; drug- or toxin-induced polyneuropathy.
* Acute demyelinating neuropathies including Guillain-Barre syndrome.
* Any other disease that could better explain the participant's signs and symptoms.
* Any history of myelopathy or evidence of central demyelination.
* Any other known autoimmune disease that, in the opinion of the investigator, would interfere with an accurate assessment of clinical symptoms of CIDP.
* Severe psychiatric disorder (such as severe depression, psychosis, bipolar disorder), history of suicide attempt, or current suicidal ideation that in the opinion of the investigator could create undue risk to the patient or could affect adherence with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate incidence, nature and severity of TEAE's | Week 14
Evaluate incidence, nature and severity of SAE's | Week 14

SECONDARY OUTCOMES:
Evaluate the efficacy of NVG-2089 in participants with CIDP | Week 14
  Treatment-naïve Participants:
  •Percentage of participants with evidence of clinical improvement (ECI) at Week 14. ECI is defined as improvement of 1 point on the adjusted Inflammatory Neuropathy Cause and Treatment (adjusted INCAT) score, or 4 points on Inflammatory Rasch-built Overall Disability Scale (I-RODS) or 8 kilopascal (kPa) on mean grip strength (dominant hand).
  Treatment-experienced Participants:
  •Percentage of participants who meet any of the following conditions:
  * Achieving ECI at Week 14
  * No worsening in adjusted INCAT between Weeks 4 and 14
  * Worsening in adjusted INCAT between Day 1 and Week 4 (and have not received rescue medication) followed by an improvement to baseline by Week 4 and maintained through Week 14

CONTACTS AND LOCATIONS:
Locations (1):
- Nuvig Site, Denton, Texas, United States

IPD SHARING:
Plan to Share IPD: No